CLINICAL TRIAL: NCT04032106
Title: A Randomized Controlled Trial of an HPV Vaccine Intervention for Young Sexual Minority Men
Brief Title: HPV Vaccine Intervention for Young Sexual Minority Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Reiter, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-19028; NCI-2019-01223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R37CA226682 (NIH)
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subject
Keywords: HPV; Men; Vaccine
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware of the research questions being tested in the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (standard HPV information) (Active Comparator): Participants receive standard information about HPV and HPV vaccine via a mobile-friendly website.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Group B (Outsmart HPV, unidirectional vaccine reminders) (Experimental): Participants receive Outsmart HPV with unidirectional vaccine reminders (i.e. reminders that do not give participants the option to respond).
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration; Behavioral: Text Message-Based Intervention
- Group C (Outsmart HPV, interactive vaccine reminders) (Experimental): Participants receive Outsmart HPV with interactive vaccine reminders (i.e. reminders that allow participants to respond).
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration; Behavioral: Text Message-Based Intervention

INTERVENTIONS:
Other: Best Practice — Receive standard information about HPV and HPV vaccine
  Other Names: standard of care; standard therapy
  Arms: Group A (standard HPV information)
Other: Informational Intervention — Receive Outsmart HPV intervention
  Arms: Group B (Outsmart HPV, unidirectional vaccine reminders); Group C (Outsmart HPV, interactive vaccine reminders)
Other: Questionnaire Administration — Ancillary studies
Behavioral: Text Message-Based Intervention — Receive unidirectional text message vaccine reminders
  Arms: Group B (Outsmart HPV, unidirectional vaccine reminders)
Behavioral: Text Message-Based Intervention — Receive interactive text message vaccine reminders
  Arms: Group C (Outsmart HPV, interactive vaccine reminders)

SUMMARY:
This phase III trial studies how well the Outsmart HPV intervention works in increasing HPV vaccine initiation and completion among young individuals who report having a history of same-sex partners, being sexually attracted to males, or identify as gay, bisexual, or queer (i.e., sexual minority males). The Outsmart HPV intervention, which is a population-targeted, individually-tailored mHealth intervention that includes vaccine reminders, may increase HPV vaccine initiation and completion among unvaccinated young sexual minority individuals.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of the Outsmart HPV intervention on increasing HPV vaccine initiation and completion.

II. Identify mediators that explain the relationship between study arm and HPV vaccine initiation and completion.

III. Determine if intervention efficacy differs across key demographic and health-related characteristics of participants.

OUTLINE: Participants are randomized to 1 of 3 groups.

GROUP A: Participants receive standard information about HPV and HPV vaccine via a mobile-friendly website.

GROUP B: Participants receive Outsmart HPV with unidirectional vaccine reminders (i.e. reminders that do not give participants the option to respond).

GROUP C: Participants receive Outsmart HPV with interactive vaccine reminders (i.e. reminders that allow participants to respond).

Participants in all study group are followed for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender male
* Ages 18-25
* Sexual minority (reports ever having oral or anal sex with a male or being sexually attracted to males; or identifies as gay, bisexual, or queer)
* Lives in the United States (US)
* Has not received any doses of HPV vaccine
* Did not participate in the pilot study
* Read English
* Able to provide informed consent (inferred by completing the screener survey and consent form)

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender male
Enrollment: 1227 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Reiter, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marshall DJ, Gower AL, Katz ML, Bauermeister JA, Shoben AB, Reiter PL. Recruitment of Young Gay, Bisexual, and Other Men Who Have Sex With Men for a Web-Based Human Papillomavirus Vaccination Intervention: Differences in Participant Characteristics and Study Engagement by Recruitment Source in a Randomized Controlled Trial. J Med Internet Res. 2025 Jan 3;27:e64668. doi: 10.2196/64668. PMID 39752644
- [Derived] Reiter PL, Gower AL, Kiss DE, Malone MA, Katz ML, Bauermeister JA, Shoben AB, Paskett ED, McRee AL. A Web-Based Human Papillomavirus Vaccination Intervention for Young Gay, Bisexual, and Other Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Feb 24;9(2):e16294. doi: 10.2196/16294. PMID 32130192
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Standard HPV Information) | Group B (Outsmart HPV, Unidirectional Vaccine Reminders) | Group C (Outsmart HPV, Interactive Vaccine Reminders)
Started | 412 | 407 | 408
Completed | 295 | 271 | 276
Not Completed | 117 | 136 | 132

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Standard HPV Information) | Group B (Outsmart HPV, Unidirectional Vaccine Reminders) | Group C (Outsmart HPV, Interactive Vaccine Reminders) | Total
Number analyzed (Participants) | 412 | 407 | 408 | 1227
Age, Customized [Count of Participants; unit: Participants]
  Ages 18-21 | 142 | 152 | 143 | 437
  Ages 22-25 | 270 | 255 | 265 | 790
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 412 | 407 | 408 | 1227
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 188 | 198 | 193 | 579
  Non-Hispanic Black | 37 | 45 | 47 | 129
  Non-Hispanic Other | 57 | 52 | 58 | 167
  Hispanic | 130 | 112 | 110 | 352
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 412 | 407 | 408 | 1227

OUTCOME MEASURES:

1. Primary Outcome: Human Papillomavirus (HPV) Vaccine Initiation and Completion
Description: Number and proportion of participants who initiate and complete the HPV vaccine series during the study period
Time Frame: Baseline up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Standard HPV Information) | Group B (Outsmart HPV, Unidirectional Vaccine Reminders) | Group C (Outsmart HPV, Interactive Vaccine Reminders)
Number analyzed (Participants) | 412 | 407 | 408
Participants
  HPV Vaccine Series Initiation: Yes | 114 | 139 | 147
  HPV Vaccine Series Initiation: No | 298 | 268 | 261
  HPV Vaccine Series Completion: Yes | 14 | 30 | 47
  HPV Vaccine Series Completion: No | 398 | 377 | 361

2. Primary Outcome: Changes in Theoretical Constructs
Description: Changes in theoretical constructs from baseline to follow-up as assessed by study surveys. Survey items developed by the study team were used to assess changes in perceived severity of HPV-related disease (possible range of -3 to 3), response efficacy of HPV vaccine (possible range of -4 to 4), and worry about getting HPV-related disease (possible range of -3 to 3). The reported numbers represent the mean change for each construct that occurred from baseline to follow-up. For each construct, a score of 0 represents no change between survey timepoints. Change scores greater than 0 indicate an increase in that construct between survey timepoints, with more positive values indicating a greater amount of change. Change scores less than 0 indicate an decrease in that construct between survey timepoints, with more negative values indicating a greater amount of change.
Time Frame: Baseline up to 9 months
Population: Participants who completed the end-of-study survey at 9 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group A (Standard HPV Information) | Group B (Outsmart HPV, Unidirectional Vaccine Reminders) | Group C (Outsmart HPV, Interactive Vaccine Reminders)
Number analyzed (Participants) | 295 | 271 | 276
Scores on a scale
  Perceived severity of HPV-related disease | -0.04 (0.74) | 0.01 (0.79) | -0.09 (0.75)
  Response efficacy of HPV vaccine | 0.41 (0.84) | 0.58 (0.88) | 0.50 (0.85)
  Worry about getting HPV-related disease | 0.63 (0.98) | 0.56 (1.05) | 0.57 (0.98)

3. Primary Outcome: Counts of Human Papillomavirus (HPV) Vaccine Initiation by Participant Characteristics
Description: Counts of human papillomavirus (HPV) vaccine initiation by demographic and health-related characteristics as assessed by study surveys
Time Frame: Baseline up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Standard HPV Information) | Group B (Outsmart HPV, Unidirectional Vaccine Reminders) | Group C (Outsmart HPV, Interactive Vaccine Reminders)
Number analyzed (Participants) | 412 | 407 | 408
Participants
  Ages 18-21 | 41 | 53 | 46
  Ages 22-25 | 73 | 86 | 101
  High school education or less | 33 | 44 | 39
  Some college education or more | 81 | 95 | 108
  Preventive health visit within the last year | 56 | 65 | 66
  No preventive health visit within the last year | 58 | 74 | 81

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Group A (Standard HPV Information) | Group B (Outsmart HPV, Unidirectional Vaccine Reminders) | Group C (Outsmart HPV, Interactive Vaccine Reminders)
All-Cause Mortality (participants affected / at risk) | 0/412 | 0/407 | 0/408
Serious Adverse Events (participants affected / at risk) | 0/412 | 0/407 | 0/408
Other Adverse Events (participants affected / at risk) | 0/412 | 0/407 | 0/408

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04032106/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04032106/ICF_002.pdf